CLINICAL TRIAL: NCT05513326
Title: Effectiveness of a 6-week Specific Rehabilitation Program Combining Education and Exercises on Walking Capacity in Patients with Lumbar Spinal Stenosis with Neurogenic Claudication
Brief Title: Effectiveness of a 6-week Specific Rehabilitation Program on Walking Capacity in Patients with Lumbar Spinal Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UQTR-2022-program
Record Dates: First submitted 2022-07-07; First posted 2022-08-24 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Spinal Stenosis
Keywords: Spinal Stenosis; Neurogenic claudication; Walking capacity; Exercises; Education; gait pattern characteristics
MeSH Terms: conditions — Spinal Stenosis; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will received education and a specific rehabilitation program (exercises).
  Interventions: Other: Exercises and education
- Control Group (Other): Control group will received education alone.
  Interventions: Other: Education alone

INTERVENTIONS:
Other: Exercises and education — Exercises: 3 training sessions per week that will last for 30 minutes. Sessions will start with 5 minutes of activation (walking on a treadmill or cycling). Then, participants will be asked to complete 5 exercises targeting lower limb strengthening (time: 18 minutes) followed by 2 exercises designed to improve balance and 3 stretching exercises for the lower limb (time: 7 minutes).
  Education: Two one-on-one sessions (during week 2 and week 4 assessments) during which participants will receive information directly related to LSS and NC using illustration and videos. Participants will also be invited to ask their questions.
  Arms: Intervention Group
Other: Education alone — Education: Two one-on-one sessions (during week 2 and week 4 assessments) during which participants will receive information directly related to LSS and NC using illustration and videos. Participants will also be invited to ask their questions.
  Arms: Control Group

SUMMARY:
The aim of this study is to determine the effectiveness of a 6-week specific rehabilitation program combining education and exercises on walking capacity in patients with LSS causing NC.

The intervention group will receive standardized education and specific exercises while the control group will only receive standardized education. The program in both groups will last for 6 weeks with 4 evaluation timepoints (baseline, week 2, week 4 and post-intervention assessment). The primary outcomes will be walking capacity measured with the Self-Paced Walking Test and the secondary outcomes will be back and leg pain intensity, LSS-related disability, self-efficacy, level of physical activity, anxiety and depression, physical activity level, gait pattern characteristics, balance, and global perceived change.

ELIGIBILITY:
Inclusion Criteria:

* being at least 50 years old
* having a degenerative central LSS alone or in combination with other LSS types (e.g. foraminal, lateral) and/or a spondylolisthesis affecting one or multiple vertebral levels, confirmed by clinical history, physical examination and proper imaging
* having NC associated with LSS
* being able to speak and understand French
* being willing to attend 3 intervention sessions per week
* with a duration of signs and symptoms of at least 3 months
* (7) being able to walk at least 20 meters without walking aid, but not being able to walk continuously for 30 minutes
* being able to provide informed written consent.

Exclusion Criteria:

* congenital LSS,
* symptomatic osteoarthritis (hip or knee) causing limited walking capacity
* neurological disease affecting walking capacity such as Parkinson
* uncontrolled diabetes
* heart failure
* intermittent claudication of vascular origin
* impaired cognitive capacity
* back or lower extremities surgery in the past 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in walking capacity | Baseline, week 2, week 4, week 6, week 12
  Walking capacity measure with the Self-Paced Walking Test (time)

SECONDARY OUTCOMES:
Change from baseline in leg and back pain intensity | Baseline, week 2, week 4, week 6, week 12
  Leg and back pain intensity will be independently assessed using a 11-point numerical rating scale (from 0 to 10 points). Higher score indicates higher pain.
Change from baseline in lumbar spinal stenosis related disabiltity | Baseline, week 6, week 12
  Lumbar spinal stenosis related disability is measured with the French-Canadian version of the Swiss Spinal Stenosis Questionnaire. Pain, function and satisfaction related to lumbar spinal stenosis. Pain subscale score range from 7 to 35 with higher values indicate a worst outcome, Function subscale score range from 5 to 20 with higher values indicate a worst outcome, Satisfaction subscale score range from 6 to 24 with higher values indicate a worst outcome. The total score is composed of the three subscales and range from 18 to 79.
Changes from baseline in self-efficacy | Baseline, week 6, week 12
  Measured with Self-efficacy measured with the French-Canadian Chronic Pain Self-Efficacy Scale. Each question is rated on a numerical scale (from 1 to 10). Total is calculated using the mean of the 33-items scores and ranges from 1 to 10 with a higher score indicate higher self-efficacy.
Change from baseline in anxiety and depression | Baseline, week 6, week 12
  Measured with the French-Canadian adaptation of the Hospital Anxiety and Depression Scale. Total score range from 0 to 21 with higher score indicating symptoms of anxiety and/or depression.
Change from baseline in physical activity level | Baseline, week 6, week 12
  Physical activity level assessed with the [Physical Activity Questionnaire for the Elderly]. The questionnaire allows to place participants into one of the 3 categories (low, moderate or high physical activity level). Physical activity level is measured in time per day.
Patient's global impression of change | changes of the global impression of change throughout the study (baseline, week 2, week 4, week 6, week 12)
  Global impression of change will be measured using a 7-point scale that ranges from 'very much improved' to 'very much worse' with 'no change' as the mid-point.
Change from baseline in biomechanical parameters of gait | Baseline, week 2, week 4, week 6, week 12
  Spatio-temporal parameters of gait measured with wearable inertial sensors (velocity (m/s))
Change from baseline in biomechanical parameters of gait | Baseline, week 2, week 4, week 6, week 12
  Spatio-temporal parameters of gait measured with wearable inertial sensors measured in meters (stride length, swing witdh, toe clearance)
Change from baseline in biomechanical parameters of gait | Baseline, week 2, week 4, week 6, week 12
  Spatio-temporal parameters of gait measured with wearable inertial sensors measured in % (walking phases, assymetry, variability)
Change from baseline in lower extremity physical function and balance | Baseline, week 6, week 12
  Lower extremity physical function and balance measured with the Short Physical Performance Battery. Total score ranges from 0 to 12 with higher score indicating a better lower extremity physical function and balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

REFERENCES:
- [Derived] Houle M, Tetreau C, Chatillon CE, Marchand AA, Descarreaux M. Effectiveness of a 6-week specific rehabilitation program combining education and exercises on walking capacity in patients with lumbar spinal stenosis with neurogenic claudication: a randomized controlled clinical trial protocol. Trials. 2022 Dec 27;23(1):1046. doi: 10.1186/s13063-022-07011-3. PMID 36572884